CLINICAL TRIAL: NCT03127280
Title: Can Investigators Reduce Urinary Catheter Use and Lower Urinary Tract Infection Among Women Undergoing Benign Gynecologic Surgery?
Acronym: CAUTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Patrick Lang, Fellow Physician, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-38
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Urinary Tract Infections; Urinary Retention; Satisfaction
Keywords: urinary tract infections; postoperative voiding dysfunction; foley removal; patient satisfaction
MeSH Terms: conditions — Urinary Tract Infections; Urinary Retention; Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Foley Care (No Intervention): Following surgery, the patient's Foley catheter is removed on the morning of post-operative day one.
- Fast Tract Foley care (Experimental): Following surgery, the patient's Foley catheter is removed on post-operative day zero, four hours after the completion of surgery.
  Interventions: Other: Fast Track foley removal

INTERVENTIONS:
Other: Fast Track foley removal — Foley catheter is removed at 4 hours after surgery
  Arms: Fast Tract Foley care

SUMMARY:
This is a randomized comparative trial investigating two different catheter management strategies among post-gynecologic surgery patients. Women undergoing any benign gynecologic surgery wherein they are anticipated to stay at least overnight and in whom no prolapse or urinary tract surgery was concurrently performed, will be randomly assigned to either conventional urinary catheter care removal on post-operative day 1 or same day surgery urinary catheter removal. Patient satisfaction and lower urinary tract symptoms including urine culture and antibiotic use will be tracked across both cohorts over the 2 weeks following the index surgery.

DETAILED DESCRIPTION:
METHODS:

This study will be conducted at The Christ Hospital. Informed consent will be obtained from the patients in the pre-operative care unit prior to administration of any medications. Candidates for the study will clearly understand consenting to enroll in the study includes not only the randomized assignment of urinary catheter care postoperatively but also a follow-up phone survey to be administered approximately 2 weeks after discharge. Patient reasons for not enrolling in the study will be recorded.

Study population All women presenting to The Christ Hospital for gynecologic surgery anticipated to require an at least 1 night stay and in whom would be expected to have an indwelling catheter overnight are eligible to participate in the study. Patients with a current urinary tract infection being treated with antibiotic(s), anticipated concomitant prolapse or incontinence surgery, a preoperative diagnosis of gynecologic malignancy, a history of chronic indwelling catheter use, a history of renal transplant or current dialysis use, or intraoperative lower urinary tract injury necessitating prolonged postoperative catheter use are to excluded from study participation. Following application of the inclusion and exclusion criteria, postoperative urinary catheter care (conventional vs. fast track) will randomized upon arrive to the postoperative care unit (PACU). These patients will compose the study population.

Protocol:

Per routine anesthesia practice once a patient has met criteria for discharge from the PACU, and following randomization into either the conventional or fast track cohorts, the subject will either have immediate removal of the catheter with a trial of void or the catheter will remain in place over night per routine practice with a trial of void arranged at the time of discharge.

The trial of void protocol will consist of backfilling the existing catheter with 300cc of sterile saline (or to a volume the patient reports to be subjectively full) and recording her voided volume that should occur within 30 minutes. The patient's self-reported percent of normal force of stream will be recorded (0-100% in 10% increments) along with her voided volume. If the patient voids at least 150cc of the instilled volume OR reports at least a >50% of normal force of stream she will be considered to have passed the voiding trial. The patient will be scanned for residual urine volume following the next spontaneous void or any time she reports symptoms consistent with obstructed voiding.

Duration of catheter use will be determined as the time from placement in the operating room (time 0) to the time it is removed on the hospital ward. Time will be recorded in hours. Discharge from the hospital will occur per the attending physician's routine practice. At hospital discharge subjects will complete a brief survey recording bladder function before and during their hospitalization. Also included in this survey will be an assessment of their overall satisfaction with their catheter management and hospital stay. Institution standard practice is to obtain a urinalysis in the operating room on all patients anticipating an overnight stay. This urinalysis and any other urine studies obtained during the hospitalization will be extracted from the medical record. The number of subjects who fail the trial of voiding between cohorts will be collected from the electronic medical record (EMR). After discharge, subjects will be contacted by phone 2-3 weeks after the index surgery. At this call subjects will be administered a survey reviewing their post-surgery bladder function including symptoms of a bladder infection. A review of the patient's hospital record will also be conducted to identify any additional urine studies ordered during the 2-3 weeks following surgery.

Randomization protocol: Permuted block randomization will be used to ensure a balanced enrollment of patients in the clinical trial. Selecting a block size of 4 will ensure that for every four patients enrolled, 2 will be assigned to the "Fast-track" cohort and 2 will be assigned to the "Conventional" cohort. In order to effectively conceal the randomization sequence, investigators will use sequentially numbered, opaque sealed envelopes (SNOSE). It will not be feasible to blind the physician, nurse and patient in this study, they will all be aware of the randomized allocation assignment. The study personnel administering the postoperative telephone questionnaires will be blinded by simply not informing them of the group allocation of the patient. Plans to manage incomplete data between cohorts will include meeting with nursing managers and supervisors to ensure that questions are completed and to verify how to enter information into the EMR. At the completion of the study every effort will be made to have all patient questionnaire completed.

ELIGIBILITY:
Inclusion Criteria:

* All women, over the age of 18, presenting to The Christ Hospital for gynecologic surgery anticipated to require an at least 1 night stay and in whom would be expected to have an indwelling catheter overnight are eligible to participate in the study.

Exclusion Criteria:

* Patients with a current urinary tract infection being treated with antibiotic(s), anticipated concomitant prolapse or incontinence surgery, a preoperative diagnosis of gynecologic malignancy, a history of chronic indwelling catheter use, a history of renal transplant or current dialysis use, or intraoperative lower urinary tract injury necessitating prolonged postoperative catheter use are to excluded from study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological females are eligible for this study as the study is only investigating patients undergoing gynecologic surgery (e.g. hysterectomy)
Enrollment: 200 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Foley Duration | Between 4 hours after surgery completion to 24 hours after surgery completion
  Determine the duration (in hours) of urinary catheter use between conventional urinary catheter care and "fast track" urinary catheter care among women undergoing benign gynecologic surgery not involving lower urinary tract surgery or pelvic organ prolapse repair.

SECONDARY OUTCOMES:
Incidence of urinary tract infection | 2-3 weeks after surgery
  Determine the number of women treated for a urinary tract infection between "conventional" urinary catheter care and "fast track" urinary catheter care over the 2 weeks following the index gynecologic surgery.
Patient satisfaction | 2-3 weeks after surgery
  Determine patient satisfaction among women exposed to conventional catheter care and "fast track" catheter care as determined by completion of a researcher designed survey, entitled "Satisfaction with Urinary Catheter management and Expectations for bladder function after discharge", prior to discharge.
Voiding dysfunction | Between 4 hours after surgery completion to 24 hours after surgery completion.
  Determine the numbers of women who fail a voiding trial between conventional catheter care and "fast track" catheter care.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lang, MD, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apisarnthanarak A, Rutjanawech S, Wichansawakun S, Ratanabunjerdkul H, Patthranitima P, Thongphubeth K, Suwannakin A, Warren DK, Fraser VJ. Initial inappropriate urinary catheters use in a tertiary-care center: incidence, risk factors, and outcomes. Am J Infect Control. 2007 Nov;35(9):594-9. doi: 10.1016/j.ajic.2006.11.007. PMID 17980238
- [Background] Umscheid CA, Mitchell MD, Doshi JA, Agarwal R, Williams K, Brennan PJ. Estimating the proportion of healthcare-associated infections that are reasonably preventable and the related mortality and costs. Infect Control Hosp Epidemiol. 2011 Feb;32(2):101-14. doi: 10.1086/657912. PMID 21460463
- [Background] Chenoweth CE, Saint S. Urinary tract infections. Infect Dis Clin North Am. 2011 Mar;25(1):103-15. doi: 10.1016/j.idc.2010.11.005. Epub 2010 Dec 18. PMID 21315996
- [Background] Saint S. Clinical and economic consequences of nosocomial catheter-related bacteriuria. Am J Infect Control. 2000 Feb;28(1):68-75. doi: 10.1016/s0196-6553(00)90015-4. PMID 10679141
- [Background] Jarvis WR. Selected aspects of the socioeconomic impact of nosocomial infections: morbidity, mortality, cost, and prevention. Infect Control Hosp Epidemiol. 1996 Aug;17(8):552-7. doi: 10.1086/647371. PMID 8875302
- [Background] Tambyah PA, Knasinski V, Maki DG. The direct costs of nosocomial catheter-associated urinary tract infection in the era of managed care. Infect Control Hosp Epidemiol. 2002 Jan;23(1):27-31. doi: 10.1086/501964. PMID 11868889
- [Background] Saint S, Veenstra DL, Lipsky BA. The clinical and economic consequences of nosocomial central venous catheter-related infection: are antimicrobial catheters useful? Infect Control Hosp Epidemiol. 2000 Jun;21(6):375-80. doi: 10.1086/501776. PMID 10879567
- [Background] Albo ME, Richter HE, Brubaker L, Norton P, Kraus SR, Zimmern PE, Chai TC, Zyczynski H, Diokno AC, Tennstedt S, Nager C, Lloyd LK, FitzGerald M, Lemack GE, Johnson HW, Leng W, Mallett V, Stoddard AM, Menefee S, Varner RE, Kenton K, Moalli P, Sirls L, Dandreo KJ, Kusek JW, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Burch colposuspension versus fascial sling to reduce urinary stress incontinence. N Engl J Med. 2007 May 24;356(21):2143-55. doi: 10.1056/NEJMoa070416. Epub 2007 May 21. PMID 17517855
- [Background] Yokoe DS, Mermel LA, Anderson DJ, Arias KM, Burstin H, Calfee DP, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Kaye KS, Klompas M, Lo E, Marschall J, Nicolle L, Pegues DA, Perl TM, Podgorny K, Saint S, Salgado CD, Weinstein RA, Wise R, Classen D. A compendium of strategies to prevent healthcare-associated infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S12-21. doi: 10.1086/591060. PMID 18840084
- [Background] Lo E, Nicolle L, Classen D, Arias KM, Podgorny K, Anderson DJ, Burstin H, Calfee DP, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Kaye KS, Klompas M, Marschall J, Mermel LA, Pegues DA, Perl TM, Saint S, Salgado CD, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent catheter-associated urinary tract infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S41-50. doi: 10.1086/591066. No abstract available. PMID 18840088
- [Background] Dziura JD, Post LA, Zhao Q, Fu Z, Peduzzi P. Strategies for dealing with missing data in clinical trials: from design to analysis. Yale J Biol Med. 2013 Sep 20;86(3):343-58. eCollection 2013 Sep. PMID 24058309
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Lang P, Quezada Y, Whiteside J. Urinary Catheter Management Approaches Among Women Undergoing Benign Gynecologic Surgery: A Randomized Trial. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):e73-e77. doi: 10.1097/SPV.0000000000000781. PMID 31688528